CLINICAL TRIAL: NCT05115305
Title: Validation of a Level 2 Sleep Study Device
Brief Title: Prodigy, a Level 2 Sleep Study Device, Validation Study
Status: Completed | Type: Observational
Sponsor: Cerebra Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: ProdigyValidationStudy
Record Dates: First submitted 2021-10-20; First posted 2021-11-10 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Sleep Apnea
Keywords: Prodigy
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Prodigy system, developed by Cerebra Medical Ltd, allows for the generation of the same information in the home that is currently only obtained in in-laboratory studies.

The objective of the current study is to demonstrate that the signals obtained by this comprehensive, portable system are comparable to those obtained in in-laboratory studies.

DETAILED DESCRIPTION:
This study consists of obtaining standard polysomnography signals concurrently by the Prodigy 2 and by the standard commercial systems used in the Sleep Disorders Clinic (Alice G3) in Hamilton, ON and the St. Charles Sleep Disorders Center (Nihon Kohden) in Port Jefferson, NY. 42 patients will be recruited from each of the two sites, for a total of 84 patients. Questionnaires on demographics and mental health, including the Depression Anxiety Stress Scale-21, questionnaires on sleep and fatigue including Pittsburgh Sleep Quality Index, Insomnia Severity Index, and Epworth Sleepiness Scale and questionnaires on quality of life including the Functional Outcomes of Sleep Questionnaire-10 (FOSQ-10) and the Euroquol 5D-5L will be completed online using a survey platform (Qualtrics or RedCap).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing a diagnostic sleep test

Exclusion Criteria:

* in-hospital patients
* subjects who self-report a previous diagnosis of neuromuscular disorders, obesity hypoventilation, or severe lung disease
* subjects who are not fluent in English, or who have special communication needs
* subjects who have dementia/Alzheimer's disease
* subjects with comorbid violent parasomnias
* subjects requiring additional assistance or who have limited ability follow commands.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients referred to either sleep clinic to undergo a diagnostic sleep test.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time | Concurrent measurement for one night
  To compare Level 1 and Level 2 sleep tests on TST
Apnea-Hypopnea Index | Concurrent measurement for one night
  To compare Level 1 and Level 2 sleep tests on AHI
Periodic Limb Movement Index | Concurrent measurement for one night
  To visually compare Level 1 and Level 2 sleep tests on PLM

SECONDARY OUTCOMES:
Signal Quality | Concurrent measurement for one night
  To compare signal quality between Level 1 and Level 2 sleep tests

CONTACTS AND LOCATIONS:
Overall Officials: Amy Bender, PhD, Principal Investigator — Cerebra Medical; Raymond Gottschalk, MD, Principal Investigator — Hamilton Sleep Disorders Clinic; Mohammad Amin, MD, Principal Investigator — St Charles Sleep Disorders Center
Locations (2):
- St Charles Sleep Disorders Center, Port Jefferson, New York, United States
- Hamilton Sleep Disorders Clinic, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Chasens ER, Ratcliffe SJ, Weaver TE. Development of the FOSQ-10: a short version of the Functional Outcomes of Sleep Questionnaire. Sleep. 2009 Jul;32(7):915-9. doi: 10.1093/sleep/32.7.915. PMID 19639754
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777